CLINICAL TRIAL: NCT05865587
Title: A QUALITATIVE RESEARCH ON THE EXPERIENCES OF PEDIATRIC EMERGENCY SERVICE PROFESSIONALS WITH REFUGEE PATIENTS
Brief Title: THE EXPERIENCES OF PROFESSIONALS WITH REFUGEE PATIENTS
Status: Withdrawn | Type: Observational
Why Stopped: Data saturation was reached when health professionals began to use similar or same expressions and it was achieved with 12 health professionals
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Mukaddes Demir Acar, Ass. Prof., Tokat Gaziosmanpasa University
Other Study IDs: TOGUMDEMIR
Record Dates: First submitted 2023-04-30; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Emergencies; Health Personnel Attitude; Child Development; Qualitative
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was conducted to examine the experiences and feelings of health professionals while providing care to refugee children and families in pediatric emergency service.

ELIGIBILITY:
Inclusion Criteria:

* Health professionals who worked in the pediatric emergency department for at least 1 year were included.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The total number of healthcare professionals working in the pediatric emergency unit is 17 [8 doctors, 9 nurses]. Health professionals who worked in the pediatric emergency department for at least 1 year were included. Two health professionals were working for less than one year and three of them were on leave. The study was completed with a total of 12 health professionals, 8 females and 4 males. Although there is no rule specified for sample size in literature for qualitative studies, situations such as the data repeating and not obtaining additional data are important indicators for terminating the application (Yıldırım & Şimşek, 2011b). Data saturation was reached when health professionals began to use similar or same expressions and it was achieved with 12 health professionals [4 doctors, 8 nurses].
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
This qualitative research data were collected by semi-structured interview form | 1 month
  In order to collect data, the researchers prepared four open-ended, basic questions: (1) What are your feelings about the refugees who migrated to our country? Can you explain? (2) Can you explain the feelings and experiences with refugee patients in pediatric emergency service? (3) How did working with refugee patients affect your thoughts about your profession? (4) What kind of problems did you experience while providing care to refugee patients in pediatric emergency services?

CONTACTS AND LOCATIONS:
Overall Officials: Selda Yüzer Alsaç, DR, Study Director — Yozgat Bozok University
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No